CLINICAL TRIAL: NCT05042154
Title: Prevalence of OSA in COPD and the Clinical Impact of OSA Diagnosis and Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Matthew Epstein, MD, Atlantic Health System
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1753461-1
Record Dates: First submitted 2021-09-08; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Prevalence of OSA in Patients Hospitalized With COPD Exacerbation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Cohort for COPD (No Intervention): Standard care patients will receive routine clinical management as per their treating physicians based on the GOLD Criteria.
- WatchPAT Cohort (Active Comparator): Consented patients will undergo group randomization to either standard AECOPD care or to the WatchPAT One cohort (WPC). The WPC will undergo a single night of in-hospital sleep apnea testing from 2200 to 0600 using the WatchPAT One, a portable and disposable home sleep apnea testing device (Itamar Medical, Israel [WPAT]).
  Interventions: Device: WatchPAT

INTERVENTIONS:
Device: WatchPAT — The WatchPAT One can detect the presence of OSA based on measurement of peripheral arterial tone (PAT), pulse rate, oxygen saturation, actigraphy, snoring, and body position.
  Arms: WatchPAT Cohort

SUMMARY:
COPD is a major cause of morbidity and mortality and is characterized by breathing impairment and related symptoms. Obstructive sleep apnea (OSA) is a highly prevalent condition that adversely affects breathing during sleep. The co-occurrence of OSA and COPD in an individual has been referred to as the overlap syndrome (OVS). Regardless of whether OVS represents a single unique entity or two separate conditions in the same patient, the combined respiratory derangements of OSA and COPD are felt to be synergistic. Patients with COPD and OSA may have more frequent and severe nocturnal arterial hypoxemia and hypercapnia than in patients with OSA alone, as well as increased pulmonary hypertension and dysrhythmias. The reported prevalence of OSA in COPD varies widely depending on patient setting, COPD severity, diagnostic methodology, etc., ranging from 10 to 75%. The presence of OSA in patients with COPD has also been implicated as a risk factor for COPD exacerbations and associated hospitalizations.

The coexistence of OSA and COPD is associated with increased risk of COPD exacerbation and shorter time to first exacerbation following diagnosis. 20% of patients discharged following an exacerbation of COPD are readmitted within 30 days, usually for respiratory-related problems.

A randomized controlled trial on Gagnon 3 at Morristown Medical Center will be conducted to diagnose OSA in patients admitted with AECOPD. The WatchPAT One device will be used and can detect the presence of OSA. If OSA is diagnosed, the patient will then be offered and prescribed a home CPAP for use after hospital discharge. We will investigate 30-day of AECOPD readmission rates.

DETAILED DESCRIPTION:
1. The initial phase of the study will be a prospective cohort design to determine the prevalence of OSA in outpatients with stable COPD who are part of the Atlantic Medical Group/ Pulmonary and Allergy Associates. Home sleep apnea testing will be performed using WatchPAT on consecutive, unselected outpatients with COPD (GOLD stage 3 or 4) who are being managed in an office setting. Inclusion criteria will include age 18 or greater, ability to participate and known dx of COPD with GOLD stage 3 or 4.
2. A second phase of our trial will determine OSA prevalence in hospitalized patients admitted with AECOPD who are part of the Atlantic Medical Group/ Pulmonary and Allergy Associates (AMG/PAA). This observational cohort will include both new admissions and 30-day readmissions. Inclusion criteria will include a primary admitting diagnosis of AECOPD, age 18 or greater, ability to participate and known dx of COPD with GOLD stage 3 or 4.
3. A third study phase will enroll COPD patients admitted to the pulmonary care unit of Morristown Medical Center and Overlook Medical Center under AMG / PAA. This phase will randomize diagnostic testing and initiate CPAP treatment in those testing positive for OSA. We will then determine CPAP treatment in those with COPD and OSA has an impact on subsequent 30-day hospital readmissions.

   Inclusion criteria for this phase of our study will include an admission diagnosis of AECOPD, age greater than 18 years, ability to participate in a portable sleep monitoring study, known COPD diagnosed by a pulmonologist (defined by GOLD, GOLD stage 3 or 4. Standard care patients will not be tested for OSA and will receive routine clinical management as per their treating physicians based on the GOLD Criteria. Consented patients will undergo group randomization to either standard AECOPD care or to overnight sleep apnea testing with the WatchPAT (Itamar Medical, Israel). If OSA is diagnosed, patients will then be offered and prescribed a home CPAP for use upon hospital discharge. The authors will investigate the percentage of 30- day acute exacerbation of COPD (AECOPD) readmission rates for both patient groups once discharged home.

   Questionnaire data will be collected from all participants regarding OSA risk factors, sleepiness, fatigue, quality of life.
4. The primary outcome is reduction in 30-day COPD hospital readmissions. Secondary outcomes include determining the prevalence of OSA in outpatient and hospitalized COPD patients. Tertiary outcomes will relate to CPAP usage and compliance, as well as other measures of sleep quality and quality of life on CPAP.

Timeline of Proposal Pre-study Months 0-6 Study Period Months 6-12 Post-study Months 12-24 IRB Submission Study Enrollment Protocol preparations Finalize Case Report Form Data collection and analysis Data analysis Training sessions for Gagnon 3 at MMC and 10 CD at OMC Ongoing clinical follow-up and management of OSA and COPD Generate hypotheses for future research studies

For the diagnostic phases of the study on out-patients and in-patients, we will include 50-100 patients' total. For the randomization portion of the study, we will include 300 patients.

Inclusion criteria include GOLD stage 3 or 4 for outpatients and for in-patients, criteria will include an admission diagnosis of AECOPD, age greater than 18 years, ability to participate in a supine sleep study, known COPD diagnosed by a pulmonologist (GOLD stage 3 or 4). Informed consent will be obtained from each patient. The study population will be composed of patients admitted to the pulmonary units at our two hospitals. All new admissions to those units will be screened daily by study personnel for enrollment using the author's inclusion and exclusions criteria. Permission to approach patients and families will be requested from the attending pulmonologist.

We will exclude patients unable or unwilling to participate in the home sleep study, medical problems or medications affecting the diagnostic accuracy/application of WatchPAT One (peripheral vascular disease, peripheral neuropathy, alpha blockade), admission to the ICU, finger deformity which prevented adequate sensor application.

Questionnaire data will be obtained directly from the patient regarding OSA risk factors, sleepiness, fatigue, and quality of life.

Patients who are not enrolled in the RCT will receive the standard of care for AECOPD based on the current GOLD Guidelines. Patients who meet inclusion criteria will be enrolled in the intervention group and spend one night wearing the WatchPAT One to determine the presence of OSA.

Consented patients will undergo group randomization to either standard AECOPD care or to the WatchPAT One cohort (WPC).

The authors will use The Pittsburgh Sleep Quality Index (PSQI, a self-rated questionnaire which assesses sleep quality and disturbances over a one-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.

The authors will use the STOP BANG questionnaire developed by Chung et al. which has been widely used as a sensitive screening tool for OSA. It is composed of both subjective and objective questions. The STOP-BANG acronym stands for: Snoring history, Tired during the day, observed stop breathing while sleep, High blood pressure, BMI more than 35 kg/m2, Age more than 50 years, Neck circumference more than 40 cm and male Gender.

Epworth Sleepiness Questionnaire measures propensity to fall asleep in eight different situations.

Fatigue severity score measures level of fatigue based on nine questions to assess severity of fatigue

Long term data will be analyzed with regard to COPD status, including hospital admissions and readmissions as well as outcomes of OSA treatment with CPAP, including morbidity and mortality and quality of life.

Our primary goal is to determine the 30-day AECOPD admission and readmission rate comparing those with and without OSA.

Additional outcomes will measure prevalence of OSA in COPD and additional outcomes effected by treatment of OSA.

Randomization method will be used using the REDCap platform.

The RNs and RTs caring for patients in the "usual AECOPD care" arm will be blinded to the WatchPAT One intervention. All subjects must have enrollment, randomization, and home sleep study with the WatchPAT One on day 4 or day 5 of hospitalization.

Participants may be withdrawn from the study without their consent if they are unable to tolerate the sleep testing or comply with other aspects of their medical care.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria include GOLD stage 3 or 4 for outpatients and for in-patients, criteria will include an admission diagnosis of AECOPD, age greater than 18 years, ability to participate in a supine sleep study, known COPD diagnosed by a pulmonologist (GOLD stage 3 or 4). Informed consent will be obtained from each patient. The study population will be composed of patients admitted to Gagnon 3 from the emergency department (ED) and to 10 CD from the ED. All new admissions to Gagnon 3 at MMC and 10 CD at OMC will be screened daily by study personnel for enrollment using the author's inclusion and exclusions criteria. Permission to approach patients and families will be requested from the attending pulmonologist.

-

Exclusion Criteria: a. List exclusion criteria:

We excluded patients unable or unwilling to participate in the home sleep study, medical problems or medications affecting the diagnostic accuracy/application of WatchPAT One (peripheral vascular disease, peripheral neuropathy, alpha blockade), admission to the ICU, finger deformity which prevented adequate sensor application.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-10-31 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
30-Day Hospitals Readmissions for COPD | 30 Days
  30-Day Hospital Readmissions from the Index COPD Hospital Stay

SECONDARY OUTCOMES:
Diagnosis of OSA | 48 hours
  Diagnosis of obstructive sleep apnea in the COPD population

IPD SHARING:
Plan to Share IPD: No